CLINICAL TRIAL: NCT02596269
Title: A Randomized Controlled Trial on the Effect and Safety of Intravenous Nefopam/Fentanyl Postoperative Patient-Controlled-Analgesia in Patients Undergoing Laparotomy
Brief Title: Nefopam/Fentanyl Postoperative Intravenous Patient-Controlled-Analgesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yong Chul Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1203-082-402
Record Dates: First submitted 2015-10-23; First posted 2015-11-04 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Laparotomy
MeSH Terms: interventions — Nefopam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nefopam(NF) group (Experimental): Received i.v. PCA with the same volume of solution containing 1250 µg fentanyl plus 120 mg of nefopam in normal saline (fentanyl 12.5 µg/ml and nefopam 1.2 mg/ml).
  Interventions: Drug: Nefopam
- Saline(SF) group (Placebo Comparator): Received i.v. PCA with 100 ml solution containing 1250 µg of fentanyl in normal saline (12.5 µg/ml),
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Nefopam — 120 mg of nefopam is included in the i.v. PCA with with 100 ml solution containing 1250 µg fentanyl. a bolus of 1 ml with an 8-min lockout time was set, without any background continuous infusion. After the end of surgery, and if the goal VRS score was achieved at PACU, PCA device was turned on and the patient was encouraged to use the pre-set bolus dose, until 24h after the end of surgery.
  Arms: Nefopam(NF) group
Drug: Saline — i.v. PCA with with 100 ml solution containing 1250 µg fentanyl. a bolus of 1 ml with an 8-min lockout time
  Arms: Saline(SF) group

SUMMARY:
BACKGROUND : There has been increasing interest on the use of nefopam in i.v. patient-controlled analgesia (PCA).

OBJECTIVE : The aim of this study was to evaluate the opioid-sparing effect of nefopam, when administered via i.v. PCA with fentanyl, after laparotomy. The adverse events associated with its use were also evaluated, and specific considerations in its clinical use were reviewed.

DESIGN : A randomized, controlled, single-centre, double-blinded study.

SETTING : One Korean university hospital.

PATIENTS : Seventy-one patients planned for elective open laparotomy

INTERVENTIONS : Patients were assigned into SF (control) or NF group, who received IV PCA with fentanyl in normal saline (25 µg/ml), or a solution with 120 mg of nefopam included (fentanyl 25 µg/ml and nefopam 1.2 mg/ml), respectively.

MAIN OUTCOME MEASURES : The pain intensity during the 24 h study period and patient satisfaction at the end of the study were evaluated. Adverse events were observed.

DETAILED DESCRIPTION:
Patients included were those planned for elective open laparotomy under general anesthesia, who were classified as American Society of Anesthesiologists (ASA) physical status I-II, with ages from 20 to 65 years.

A computer-generated randomization table was used to allocate patients equally into two groups, saline-fentanyl (SF) group (n=36) and Nefopam-fentanyl (NF) group (n=36). SF group, the control group received i.v. PCA with 100 ml solution containing 1250 µg of fentanyl in normal saline (12.5 µg/ml), while NF group, received i.v. PCA with the same volume of solution containing 1250 µg fentanyl plus 120 mg of nefopam in normal saline (fentanyl 12.5 µg/ml and nefopam 1.2 mg/ml). For both groups, a bolus of 1 ml with an 8-min lockout time was set, without any background continuous infusion during the study period.

After the end of surgery, as soon as the patient was awake, the pain intensity was assessed using the 4-points verbal rating scale (VRS) score (0: no pain, 1: mild pain, 2: moderate pain, and 3: intense pain), at 5-min interval, while staying at PACU. The pain was assessed at rest (VRS-R). If the patient reported VRS-R ≥ 3, an anesthetist not involved in the study administered a rescue dose of IV fentanyl 1 µg/kg. Then, pain was assessed every 5 min, and fentanyl given until VRS-R < 3. If the score did not fall below 3 despite 5 times of bolus fentanyl administration (30 min after arrival on PACU), the patient was dropped out of the study.

If the goal VRS score was achieved, PCA device was turned on and the patient was encouraged to use the pre-set bolus doses.

After the 30 min stay at PACU, the patients were transferred to the ward, and both numeric rating scale (NRS) pain score at rest (NRS-R) and on coughing (NRS-C) using an NRS (0-10), were recorded at 1h, 2h, 6h, 12h and 24h postoperatively. The data of cumulative PCA dose and the number of bolus doses, as displayed on the PCA device, were recorded and transferred to a computer for interpretation. No additional analgesics, antipyretics, or anti-inflammatory drug were allowed during the study.

ELIGIBILITY:
Inclusion Criteria:

* those planned for elective open laparotomy under general anesthesia, who were classified as ASA physical status I-II

Exclusion Criteria:

* the presence of renal and hepatic disease, high risk of urinary retention, seizure history, known allergy to any of the medications used, current history of psychiatric disorder, or those presently taking psychotropic medications or monoamine oxidase inhibitors.
* Patients who could not understand verbal rating scale (VRS) and 11-points numeric rating scale (NRS) pain scores, or did not sign on informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
fentanyl consumption | during the stay at PACU, at the end of intervention (24h after surgery)

SECONDARY OUTCOMES:
pain intensity (NRS scores) | 1h, 2h, 6h, 12h and 24h postoperatively
Satisfaction on analgesia using 4-points VRS (0: no satisfaction, 1: mild satisfaction, 2: moderate satisfaction, and 3: intense satisfaction) | at the end of the study (24 h after the surgery)
hypertension, tachycardia, sweating, shivering, nausea, vomiting, sedation, pruritis and/or dry mouth | Throughout study on report-based (24h)
hypertension, tachycardia | 1h, 2h, 6h, 12h and 24h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chul Kim, MD., PhD., Principal Investigator — Seoul National University Hospital, Korea

REFERENCES:
- [Background] Oh CS, Jung E, Lee SJ, Kim SH. Effect of nefopam- versus fentanyl-based patient-controlled analgesia on postoperative nausea and vomiting in patients undergoing gynecological laparoscopic surgery: a prospective double-blind randomized controlled trial. Curr Med Res Opin. 2015 Aug;31(8):1599-607. doi: 10.1185/03007995.2015.1058251. Epub 2015 Jul 9. PMID 26047392
- [Derived] Jin HS, Kim YC, Yoo Y, Lee C, Cho CW, Kim WJ. Opioid sparing effect and safety of nefopam in patient controlled analgesia after laparotomy: A randomized, double blind study. J Int Med Res. 2016 Aug;44(4):844-54. doi: 10.1177/0300060516650783. Epub 2016 Jun 29. PMID 27358262